CLINICAL TRIAL: NCT01556698
Title: Single-Center, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Comparison, Proof of Concept Study Comparing the Tolerability, Safety and Efficacy of NVN1000 Topical Gel Gel Vehicle in the Treatment of Moderate to Severe Acne
Brief Title: Study of NVN1000 Topical Gel and Topical Gel Vehicle in the Treatment of Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AC001
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Acne Vulgaris; Acne
Keywords: Acne Vulgaris; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NVN1000 Gel (Experimental): NVN1000 Gel topically applied one daily at bedtime for 8 weeks
  Interventions: Drug: NVN1000
- Vehicle Gel (Placebo Comparator): Vehicle Gel topically applied once daily at bedtime for 8 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: NVN1000
  Other Names: Nitric Oxide 0.3%
  Arms: NVN1000 Gel
Drug: Vehicle — Placebo
  Other Names: Vehicle Comparator
  Arms: Vehicle Gel

SUMMARY:
The primary objective of this study is to compare the tolerability, safety and efficacy of NVN1000 Topical Gel and Topical Gel Vehicle in the treatment of subjects with moderate to severe acne vulgaris.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the tolerability, safety and efficacy of once daily application of NVN1000 Topical Gel for 8 weeks in comparison with its vehicle in subjects with moderate to severe acne.

ELIGIBILITY:
Inclusion Criteria:

* Baseline IGA score of moderate (3) or severe (4)
* Minimum of 20 but no more than 40 facial inflammatory lesions
* Minimum of 20 but not more than 60 facial non-inflammatory lesions
* No more than 2 facial nodules

Exclusion Criteria:

* Dermatological conditions on the face that could interfere with clinical evaluations
* Underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive
* History of experiencing significant burning or stinging when applying any facial treatment
* Female subjects, if they are pregnant,nursing mothers, or planning to become pregnant during the study
* Have used estrogens or oral contraceptives for less than 90 days immediately preceding the Baseline visit, discontinued use of estrogens or oral contraceptives less than 90 days prior to Baseline,or planning to begin or discontinue use of this therapy during the treatment period
* Have used medications and/or vitamins which are reported to exacerbate acne during the 180 days immediately preceding the Baseline visit
* Use concomitantly over-the-counter (OTC) products that contain ingredients such as benzoyl peroxide,salicylic acid,alpha-hydroxy acid,retinol or glycolic acids
* Have not undergone the specified washouts for topical preparations,systemic medications and procedures noted in the protocol

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Blanco, MD, Principal Investigator — Instituto Dermatológico
Locations (1):
- Instituto Dermatologico, Santo Domingo, Dominican Republic